CLINICAL TRIAL: NCT03441607
Title: Safety & Efficacy of Micronized Human Amnion Chorion Membrane Biologic (mHACMb) FloGraft (Micronized Human Amnion Chorion Membrane)® in Adults With Pain Due to Osteoarthritis of the Knee
Brief Title: Safety & Efficacy FloGraft (Micronized Human Amnion Chorion Membrane)® in Adults With Pain Due to OA of the Knee
Acronym: OA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Applied Biologics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BX001
Record Dates: First submitted 2018-02-07; First posted 2018-02-22 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug (Active Comparator): Intervention: 40 mg of micronized human amnion chorion membrane biologic (mHACMb); administered 1(x) on second visit; followed by 2 follow-up visits for assessment over a duration of 3 months.
  Interventions: Drug: mHACMb
- Placebo (Placebo Comparator): Intervention: 1cc of saline will be administered as a one time injection on visit 2, administered 1(x) on first visit; followed by 2 follow-up visits for assessment over a duration of 3 months.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: mHACMb — Active ingredient
  Other Names: 40mg FloGraft (micronized human amnion chorion membrane)®; 100mg FloGraft (micronized human amnion chorion membrane)®
  Arms: Drug
Other: placebo — inactive ingredient
  Other Names: saline
  Arms: Placebo

SUMMARY:
Safety & Efficacy of FloGraft (Micronized Human Amnion Chorion Membrane)® in Adults With Pain Due to Osteoarthritis of the Knee.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent to participate in the study.
* Willing and able to participate in all procedures and follow-up evaluations necessary to complete the study.
* Subject is 30 years or older.
* Moderate OA pain (rating of at least 20mm on the VAS) assessed at Baseline.
* Moderate to moderately-severe OA pain in the index knee (rating of at least 1.5 on the WOMAC Index 3.1 5-point Likert Pain Subscale) assessed at Baseline.
* Must be ambulatory.
* No analgesia (including acetaminophen [paracetamol]) taken 12 hours prior to an efficacy measure.

Exclusion Criteria:

* Subject has active infection at the injection site.
* Subject has rheumatoid arthritis, psoriatic arthritis, or have been diagnosed with any other auto-immune disorders that could be the cause of their knee pain.
* BMI greater than 40 kg/m2.
* Subject has received an intra-articular hyaluronic acid (HA) injection for the treatment of OA of the target knee within 3 months prior to screening.
* Subject has received an intra-articular amniotic fluid, amniotic membrane or amniotic fluid/membrane combination injection for the treatment of OA of the target knee within 3 months prior to screening.
* Subject has received a steroid, bone marrow aspirate concentrate (BMAC) or platelet rich plasma (PRP) injection for the treatment of OA of the target knee within 3 months prior to screening.
* Subject has had major surgery, arthroplasty or arthroscopy in the target knee within 26 weeks of treatment or plans to have surgery in the target knee within 180 days of treatment.
* Subject is pregnant or plans to become pregnant within 180 days of treatment.
* Subject has used an investigational drug, device or biologic within 12 weeks prior to treatment.
* Subject has any significant medical condition that, in the opinion of the Investigator, would interfere with protocol evaluation and participation.
* Subject is currently taking anticoagulant therapy (excluding Plavix or Aspirin).
* Diagnosis of gout in the past 6 month.
* Major injury to the target knee within the 12 months prior to the screening.
* Severe hip osteoarthritis ipsilateral to the target knee.
* Any pain that could interfere with the assessment of the target knee pain (e.g. pain in any other part of the lower extremities, pain radiating to the knee).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 3 Months
  Decreased Pain Level

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC®) osteoarthritis Index 3.1. | 3 Months
  Decrease in pain, stiffness, and physical functioning of the joints.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Britt, Study Director — Applied Biologics, LLC
Locations (1):
- Texas Orthopedic Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No